CLINICAL TRIAL: NCT04589520
Title: The Effects of the App HeartBot on the Stress and Emotional Well-Being Over a 21-day Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranjani Iyer (Other)
Responsible Party: Sponsor-Investigator, Ranjani Iyer, Director of Heartfulness Program for Schools, Heartfulness Institute
Organization: Heartfulness Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019/07/11
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stress; Mental Health Wellness 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeartBot Group (Experimental): The HeartBot group downloaded the app and used it daily for 21 days based on a calendar that provided them with step by step outlines of the tools for each day.
  Interventions: Behavioral: HeartBot App
- Control Group (No Intervention): The control group did not download the app and experienced no change to their daily routines.

INTERVENTIONS:
Behavioral: HeartBot App — HeartBot is an app designed to enable people 14 years and older to use relaxation tools offered by Heartfulness to deal with daily stress and anxiety in a healthy, productive manner.
  Arms: HeartBot Group

SUMMARY:
HeartBot is an app designed to enable people 14 years and older to use relaxation tools offered by Heartfulness. The study is conducted to examine the effect of the app on stress and emotional wellness in participants 14 years and older.

Research Question: Does HeartBot affect the stress levels and emotional wellness in participants 14 years and older?

Hypothesis: Participants who use HeartBot for 21 days will see a significant decrease in their stress levels and an improvement in emotional wellness.

ELIGIBILITY:
Inclusion Criteria:

* Participants 14 years of age and older willing to participate in the study; parental/guardian consent in case of the student below 18 years of age.

Exclusion Criteria:

* Individuals less than 14 years of age. As the app is available on iOS only, you need to have an iOS device to participate.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-08-18 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Stress Levels | 21 days for 30 minutes every day based on a 21-day calendar
  Participant stress levels were measured using the Perceived Stress Scale (PSS). This 10-item scale measures the degree to which a situation in someone's life is considered stressful .

SECONDARY OUTCOMES:
Change in Emotional Wellbeing | 21 days for 30 minutes every day based on a 21-day calendar
  The emotional wellness of the participants was measured using the EPOCH measure of adolescent wellbeing. This is a 20-item scale used to measure five different positive characteristics: Engagement, Perseverance, Optimism, Connectedness, and Happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjani B Iyer, PhD, Principal Investigator — Heartfulness Institute
Locations (1):
- Ranjani B Iyer, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publish a research paper with details on the study design, protocol, analysis of data, and report on implications to stress management and wellness tools.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting six months after publication
Access Criteria: Access criteria IPD and any additional supporting information will be shared with the researchers furthering research in stress management and emotional wellness tools.

REFERENCES:
- [Derived] Iyer L, Iyer RB, Kumar V. A Relaxation App (HeartBot) for Stress and Emotional Well-Being Over a 21-Day Challenge: Randomized Survey Study. JMIR Form Res. 2021 Jan 29;5(1):e22041. doi: 10.2196/22041. PMID 33455902